CLINICAL TRIAL: NCT05726929
Title: Algology in Oncology Osteopathic Support
Brief Title: Algology in Oncology Osteopathic Support (ALGOS)
Acronym: ALGOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Toulousain d'Ostéopathie (Other)
Collaborators: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCB: 2022-A01349-34
Record Dates: First submitted 2023-01-12; First posted 2023-02-14 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Neuropathic Pain
Keywords: Supportive care; Osteopathy
MeSH Terms: conditions — Breast Neoplasms; Neuralgia | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteopathic treatment (OT) (Experimental): Osteopathic treatment, 3 sessions of 1h + Treatment As Usual (TAU)
  Interventions: Other: Osteopathic treatment; Other: Capsaicin QUTENZA Patch (TAU)
- Treatment As Usual (TAU) (Active Comparator): Treatment As Usual, Capsaicin Qutenza Patch (Conventionnal Treatment in algology in supportive care)
  Interventions: Other: Capsaicin QUTENZA Patch (TAU)

INTERVENTIONS:
Other: Osteopathic treatment — Osteopathic Manual Treatment
  Arms: Osteopathic treatment (OT)
Other: Capsaicin QUTENZA Patch (TAU) — Capsaicin QUTENZA Patch is the treatment as usual (TAU) delivered in the medical algology service

SUMMARY:
The aim of the study is to evaluate the Impact of add-on osteopathic treatment in the algological course of patients treated for breast cancer : Randomized Controlled Trial.

DETAILED DESCRIPTION:
Background: In women, the breast is the most common cancer site in the world and is unfortunately the one with the highest number of deaths. It is estimated that 30-50% of women who have undergone a mastectomy are affected by this post-operative syndrome and that 50% of patients would report chronic pain one year after surgery. Chronic pain after breast surgery (incidence of 30% at 3 months) has an essentially neuropathic component. There are many contributing factors, depending on the surgery, the patient, the analgesia technique and the treatments associated with the cancer.

Methods: The ALGOS study has received a favourable opinion from the Ethical Committee (CPP). Capsaicin patch (Qutenza 179mg) treatment as usual (TAU) is delivered in medical algological care in Oncopole, Toulouse, France. In total 120 patients meeting the inclusion criteria will be randomly assigned to one of the 3 treatment groups: One receiving osteopathic treatment before the TAU (Group 1) ; The second group receiving the OT in addition to and during the TAU (Group 2) ; The third group will receive OT after the TAU and if considered in "therapeutic failure" (Group 3). Each group will have his own control (G1C-G2C-G3C). All the patients in group 1,2,3 will receive 3 1-hour osteopathic treatment sessions in a "backbox" strategy of treatment.

The TAU by Qutenza is defined and recommended by the French health high authority. The primary outcome is the evaluation of neuropathic pain by DN4 score. The secondary outcomes include superficial fascial tissue properties of the scar by MyotonPRO, the therapeutic alliance quality will be evaluated by the Working Alliance Inventory (WAI) and the impact of pain in their quality of life by the Brief Pain Inventory (BPI score).

Discussion: If the results of the ALGOS study are positive, the study will provide arguments in favor of osteopathic treatment as a possible non-invasive additional treatment option in the multidisciplinary care support approach for patients with neuropathic pain after a breast cancer.

Trial Registration: Date: Release December-09, 2022 (positive opinion from ethical committee CPP) /N° ID-RCB: 2022-A01349-34.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with sequelae of pain following breast cancer surgery with or without other treatments and who have been in pain for more than 3 months. Neuropathic pain may be experienced in the upper and middle chest, armpit and/or arm ipsilateral to the surgery and/or radiotherapy.

Exclusion Criteria:

* Unemancipated minors, protected adults and adults who are not in a position to give their consent are excluded from the protocol.
* Patients who do not have social security coverage
* Patients with non-iatrogenic peripheral neuropathy
* Patients who do not speak French
* Patients with confusional disorders
* Patients with a brain tumour
* Any patient with healing disorders at the surgical site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
Changes in Neuropathic pain assessment from baseline to 9 months | 5 minutes of test / Day 0 (inclusion) / every 3 months / at the end of the study 9 months after inclusion
  Neuropathic pain assessment in 4 points (DN4 questionnaire) 10 questions / A result more than 4/10 means a neuropathic pain component. 0 = minimum 10 = maximum

SECONDARY OUTCOMES:
Changes in Brief Pain Inventory from baseline to 9 months | 10 minutes / Evaluation Every 3 months and at the end of the study after 9 months
  Impact of pain in the quality of life (Brief Pain Inventory Score) / 9 questions with scales 0 to 10, where 0 = No pain and 10 = Maximal pain or impact
Changes in Viscoelastic Scar Tissue Properties from baseline to 9 months | 5 minutes of measurements / Day 0 at inclusion and at each Osteopathic session every 15days (3 sessions) and at the end of the study 9 months after inclusion.
  Mechanical Fascial tissue properties evaluated by MyotonPRO device (Validity/reliability confirmed in scientific research). This is a Non invasive device. A standardized force ( 0.48N) applied on the superficial skin to study the mechanical oscillation in response of the deformation. Variables measured are the Tone (Hz), Stiffness (N/m), Logaryhmic decrement, Relaxation time (ms). All these parameters traduce the "state of tone -elasticity" of the fascial tissue. (Higher is the stiffness value higher is the state of tone. Lower is the value lower is the tension).

OTHER OUTCOMES:
Working Alliance Inventory | 10 minutes / evaluation at the end of Osteopathic consultation n°2 at 1.5 month.
  Score to evaluate the quality of therapeutic alliance / 36 questions each item is scored from 1 (minimum) to 7 (maximum) / Global score on 252 / Higher scores reflects a more positive rating of working alliance

CONTACTS AND LOCATIONS:
Overall Officials: Loïc TREFFEL, PhD, Principal Investigator — Institut Toulousain d'Ostéopathie
Locations (1):
- Institut Claudius Regaud Toulouse Oncopole, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided